CLINICAL TRIAL: NCT06605235
Title: The Ideal Local Anesthetic for Intraperitoneal Gallbladder Bed Infiltration Following Laparoscopic Cholecystectomy - a Randomized Controlled Trial
Brief Title: The Ideal Local Anesthetic for Intraperitoneal Gallbladder Bed Infiltration Following Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Air Force (PAF) Hospital Islamabad (Other)
Responsible Party: Principal Investigator, Syed Moiz Ahmed, Post-graduate resident, Principle Investigator, Department of General Surgery, Pakistan Air Force (PAF) Hospital Islamabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SGR-2021-137-2499-1; SGR-2021-137-2499-1 (Other: PAF Hospital ethical committee)
Record Dates: First submitted 2024-09-14; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cholecystectomy, Laparoscopic; Pain Management
Keywords: laparoscopic cholecystectomy; lignocaine; bupivacaine; visual analogue scale
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lignocaine (Experimental): patients received 20 ml of 1% lignocaine (Xyloaid-lignocaine HCl injection) infiltrated in the gall bladder bed after removal of the gall bladder, along with 10 ml of 1% lignocaine infiltration at the port sites at the end of the procedure
  Interventions: Procedure: Local Anesthesia
- Bupivacaine (Experimental): Subjects received 20 ml of 0.25% bupivacaine (Bupicain-Bupivacaine HCl injection) infiltration in gall bladder bed, along with 10 ml of 0.25% bupivacaine at port sites
  Interventions: Procedure: Local Anesthesia
- Lignocaine + Bupivacaine (Experimental): patients received 10 ml of 1% lignocaine along with 10 ml of 0.25% bupivacaine infiltrated in gall bladder bed, and then 5 ml of 1% lignocaine along with 5 ml of 0.25% bupivacaine at the port sites
  Interventions: Procedure: Local Anesthesia

INTERVENTIONS:
Procedure: Local Anesthesia — In Group A, patients received 20 ml of 1% lignocaine (Xyloaid-lignocaine HCl injection) infiltrated in the gall bladder bed after removal of the gall bladder, along with 10 ml of 1% lignocaine infiltration at the port sites at the end of the procedure. Subjects in Group B received 20 ml of 0.25% bupivacaine (Bupicain-Bupivacaine HCl injection) infiltration in gall bladder bed, along with 10 ml of 0.25% bupivacaine at port sites. In Group C patients received 10 ml of 1% lignocaine along with 10 ml of 0.25% bupivacaine infiltrated in gall bladder bed, and then 5 ml of 1% lignocaine along with 5 ml of 0.25% bupivacaine at the port sites

SUMMARY:
To control pain after surgery for removal of gallbladder, local anesthetic agent can be sprayed on the liver bed from where the gallbladder is removed. This study was conducted to identify the ideal local anesthetic agent for this purpose.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the gold standard operation for symptomatic cholelithiasis; however, pain remains a major factor increasing morbidity and length of hospital stay. Infiltration of gallbladder bed with local anesthetic has been shown to improve post-operative pain after laparoscopic cholecystectomy, although, it is unclear which local anesthetic provides superior pain relief. Patients undergoing laparoscopic cholecystectomies were randomized into 3 groups of 30 patients each depending on the local anesthetic instilled in the gallbladder bed; lignocaine (Group A), bupivacaine (Group B), or a combination of lignocaine and bupivacaine (Group C). Pain was measured using visual analogue score at 2-, 6-, 12- and 24-hours following surgery

ELIGIBILITY:
Inclusion Criteria:

* elective/emergency laparoscopic cholecystectomy
* ASA grade I/II
* Ages 18-75 years

Exclusion Criteria:

* patients on chronic analgesics
* pts receiving analgesics 24 hours prior to surgery
* intraoperative bile spillage or drain placement
* CBD exploration or T-tube insertion
* BMI > 40 kg/m2
* pts allergic to, or otherwise not able to receive medications being tested

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale - pain score | 2-, 6-, 12-, 24-hours following surgery
  Visual analogue score to quantify pain following laparoscopic cholecystectomy. Maximum value is 10 (which means worst pain), and minimum value is 0 (which means no pain).

SECONDARY OUTCOMES:
Shoulder tip pain | within 24 hours following surgery
  The time following surgery when shoulder tip pain was gone
Flatus | within 24 hours following surgery
  Time to passing flatus
nausea/vomiting | within 24 hours following surgery
  time when nausea/vomiting was not present in the patient
Time to ambulation | within 24 hours following surgery
  time after surgery when the patient started ambulating
rescue analgesia | within 24 hours following surgery
  number of times rescue analgesia was used
Mean arterial pressure | 2-, 6-, 12-, 24-hours following surgery
  systolic and diastolic blood pressures were measured for the patients at intervals, and then mean arterial pressures were calculated
Heart rate | 2-, 6-, 12-, 24 hours
  Heart rate was measured at intervals in beats per minute
oxygen saturation | 2-, 6-, 12-, 24 hours
  oxygen saturation was noted at intervals

CONTACTS AND LOCATIONS:
Locations (1):
- PAF hospital, Islamabad, Capital Territory, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeh CN, Tsai CY, Cheng CT, Wang SY, Liu YY, Chiang KC, Hsieh FJ, Lin CC, Jan YY, Chen MF. Pain relief from combined wound and intraperitoneal local anesthesia for patients who undergo laparoscopic cholecystectomy. BMC Surg. 2014 May 12;14:28. doi: 10.1186/1471-2482-14-28. PMID 24886449
- [Background] Protic M, Veljkovic R, Bilchik AJ, Popovic A, Kresoja M, Nissan A, Avital I, Stojadinovic A. Prospective randomized controlled trial comparing standard analgesia with combined intra-operative cystic plate and port-site local anesthesia for post-operative pain management in elective laparoscopic cholecystectomy. Surg Endosc. 2017 Feb;31(2):704-713. doi: 10.1007/s00464-016-5024-5. Epub 2016 Jun 20. PMID 27324337
- [Background] Inan A, Sen M, Dener C. Local anesthesia use for laparoscopic cholecystectomy. World J Surg. 2004 Aug;28(8):741-4. doi: 10.1007/s00268-004-7350-3. Epub 2004 Aug 3. PMID 15457350
- [Background] Donatsky AM, Bjerrum F, Gogenur I. Intraperitoneal instillation of saline and local anesthesia for prevention of shoulder pain after laparoscopic cholecystectomy: a systematic review. Surg Endosc. 2013 Jul;27(7):2283-92. doi: 10.1007/s00464-012-2760-z. Epub 2013 Jan 26. PMID 23355159
- [Background] Boddy AP, Mehta S, Rhodes M. The effect of intraperitoneal local anesthesia in laparoscopic cholecystectomy: a systematic review and meta-analysis. Anesth Analg. 2006 Sep;103(3):682-8. doi: 10.1213/01.ane.0000226268.06279.5a. PMID 16931681
- [Background] Ejlersen E, Andersen HB, Eliasen K, Mogensen T. A comparison between preincisional and postincisional lidocaine infiltration and postoperative pain. Anesth Analg. 1992 Apr;74(4):495-8. doi: 10.1213/00000539-199204000-00004. PMID 1482431
- [Background] Ng A, Swami A, Smith G, Robertson G, Lloyd DM. Is intraperitoneal levobupivacaine with epinephrine useful for analgesia following laparoscopic cholecystectomy? A randomized controlled trial. Eur J Anaesthesiol. 2004 Aug;21(8):653-7. doi: 10.1017/s0265021504008117. PMID 15473621
- [Background] Rutherford D, Massie EM, Worsley C, Wilson MS. Intraperitoneal local anaesthetic instillation versus no intraperitoneal local anaesthetic instillation for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD007337. doi: 10.1002/14651858.CD007337.pub4. PMID 34693999
- [Background] Strasberg SM, Clavien PA. Overview of therapeutic modalities for the treatment of gallstone diseases. Am J Surg. 1993 Apr;165(4):420-6. doi: 10.1016/s0002-9610(05)80933-x. PMID 8480874
- [Background] Rance, G. and A. Jones, Gallstone disease. InnovAiT, 2016. 9(1): p. 7.
- [Background] Stinton LM, Myers RP, Shaffer EA. Epidemiology of gallstones. Gastroenterol Clin North Am. 2010 Jun;39(2):157-69, vii. doi: 10.1016/j.gtc.2010.02.003. PMID 20478480